CLINICAL TRIAL: NCT01904734
Title: A Comparison of Clomiphene Citrate Responses in Men With Hypothalamic Hypogonadism naïve to, and Previously Treated With, Testosterone
Brief Title: Clomid in Men With Low Testosterone With and Without Prior Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sherman M. Harman, Chief, Endocrine Division, Dept. of Internal Medicine, Phoenix VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VETSCLOMIDPHX
Record Dates: First submitted 2013-07-15; First posted 2013-07-22 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hypogonadism, Male
Keywords: testosterone; hypogonadism; pituitary
MeSH Terms: conditions — Eunuchism; Hypogonadism; Pituitary Diseases | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No previous male hormone treatment (Active Comparator): Clomiphene
  Interventions: Drug: Clomiphene
- Previously treated with testosterone (Active Comparator): Clomiphene
  Interventions: Drug: Clomiphene

INTERVENTIONS:
Drug: Clomiphene — Start with 25 mg and escalate to 50 mg in men not achieving goal for serum testosterone after 3 weeks
  Other Names: Clomid; Clomiphene citrate

SUMMARY:
This study aims to explore whether men with low testosterone levels, due to altered brain regulation of male hormone function, who have been previously treated with testosterone, respond as well as men who have not been so treated to clomiphene citrate, an agent commonly used for female infertility that has been shown to improve male hormone secretion in some cases.

DETAILED DESCRIPTION:
Clomiphene, an oral FDA-approved agent for female infertility has been shown to normalize testosterone levels in men with hypogonadotropic hypogonadism. It appears to be safe and well tolerated. This study will compare testosterone responses to clomiphene citrate in male veterans with hypothalamic hypogonadism naïve to treatment with responses of similar patients already receiving treatment with injectable or transdermal testosterone. This is an open-label, prospective, interventional trial to be conducted in an outpatient specialty care setting. We will randomize 64 hypogonadal male veterans evenly divided between naive and previous treatment and treat for 8 weeks with clomid, increasing the initial dose of 25 mg to 50 mg/day in those who fail to achieve target testosterone level (450 ng/dl) after the first 3 weeks. Endpoint measurements performed in the Phoenix VA Health Care System (PVAHCS) clinical laboratory will be total testosterone as well as bioavailable testosterone and sex hormone binding globulin. Total testosterone level at 8 weeks of treatment will be reported as the primary endpoint. Safety measures (CBC,liver functions, PSA) will be assessed at 8 weeks as well. This study will help serve as a guide for design of future studies of clomiphene in hypogonadal men.

ELIGIBILITY:
Inclusion Criteria:

* Patient or eligible for care at Phoenix VA Health Care System
* Male ages 30-70 years
* testosterone level below 250 ng/dl before treatment
* able to provide informed written consent

Exclusion Criteria:

* evidence of pituitary tumor >1mm by MRI or CAT scan
* chronic illness (renal, cardiac, liver failure)
* Prostate specific antigen (PSA) >4.0 ng/ml
* history of prostate, breast, or testicular cancer
* eye disease compromising vision (e.g. cataracts)

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Total serum testosterone | at the end of 8 weeks of treatment
  laboratory measurement by standard immunometric method

SECONDARY OUTCOMES:
Bioavailable testosterone | at the end of 8 weeks of treatment
  Non-SHBG bound testosterone by ammonium sulfate precipitation method
Serum sex hormone binding globulin (SHBG)level | at the end of 8 weeks of treatment
  Laboratory measurement of SHBG by standard immunometric technique

CONTACTS AND LOCATIONS:
Overall Officials: Sherman M Harman, MD, PhD, Principal Investigator — Phoenix VA Health Care System
Locations (1):
- Phoenix VA Health Care System, Phoenix, Arizona, United States

REFERENCES:
- [Background] Moskovic DJ, Katz DJ, Akhavan A, Park K, Mulhall JP. Clomiphene citrate is safe and effective for long-term management of hypogonadism. BJU Int. 2012 Nov;110(10):1524-8. doi: 10.1111/j.1464-410X.2012.10968.x. Epub 2012 Mar 28. PMID 22458540
- [Background] Katz DJ, Nabulsi O, Tal R, Mulhall JP. Outcomes of clomiphene citrate treatment in young hypogonadal men. BJU Int. 2012 Aug;110(4):573-8. doi: 10.1111/j.1464-410X.2011.10702.x. Epub 2011 Nov 1. PMID 22044663
- [Background] Taylor F, Levine L. Clomiphene citrate and testosterone gel replacement therapy for male hypogonadism: efficacy and treatment cost. J Sex Med. 2010 Jan;7(1 Pt 1):269-76. doi: 10.1111/j.1743-6109.2009.01454.x. Epub 2009 Aug 17. PMID 19694928